CLINICAL TRIAL: NCT00705796
Title: Influence on Human Male Fertility of Testosterone After Intranasal (MPP10) or Transdermal (AndroGel™) Application
Brief Title: Influence of Administration Route of Testosterone on Male Fertility
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: financial constraints
Sponsor: Acerus Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor, CEO U. Mattern, M et P Pharma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nasobol 02/2008
Record Dates: First submitted 2008-06-25; First posted 2008-06-26 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Hypogonadism
Keywords: Hypogonadism; Spermatogenesis; Quality of Life
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Group 1 will be treated with MPP10, 7.6 mg, twice daily to be taken immediately after waking up and washing/showering (approx. 7:00-8:00 AM) and at lunch time (approx. 12:00 AM).
  Interventions: Drug: MPP10, testosterone
- Group 2 (Active Comparator): Group 2 will be treated with AndroGel® 50 mg, once daily in the morning after washing/showering.
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: MPP10, testosterone — Testosterone intranasal, 7.6 mg, twice daily to be taken immediately after waking up and washing/showering (approx. 7:00-8:00 AM) and at lunch time (approx. 12:00 AM).
  Other Names: Nasobol
  Arms: Group 1
Drug: Testosterone — AndroGel® 50 mg, once daily in the morning after washing/showering.
  Other Names: AndroGel
  Arms: Group 2

SUMMARY:
Exogenously administered testosterone will override the normal negative feedback of endogenous testosterone on the hypothalamus and pituitary. Constantly, relatively high and constant testosterone levels will cause a drop in FSH and LH production by the pituitary. Since FSH and LH are signalling hormones to the testes, endogenous testosterone production and spermatogenesis will be down-regulated. It is expected that intranasal dosing in the morning will mimic the normal physiological pattern of testosterone production thereby avoiding negative side-effects on spermatogenesis. Trans-dermal gels give testosterone levels more or less constant over the day and will very likely have inhibitory effects on spermatogenesis.

The main objective of this study is to show that twice daily intranasal dosing does not have, or has a smaller inhibitory effect on spermatogenesis in comparison to transdermal testosterone gels.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 50 years but not older than 80 years of age;
* Serum testosterone level <13.8 nmol/l;
* Sperm concentration > 40 Million/ml;
* Willing to give written informed consent.

Exclusion Criteria:

* Testicular diseases or having had any surgical procedures applied to the testes;
* History or currently existing serious disease of any type, in particular liver, kidney or heart disease, any form of diabetes mellitus, cancer or psychiatric illness;
* Current androgen, anabolic steroid or sex hormone treatment or any treatment with such compounds in the previous 6 months;
* Blood donation within the 12-week period before the initial study dose.
* History of, or current nasal disorders (e.g. seasonal or perennial allergic rhinitis, atrophic rhinitis, polyposis, abuse of nasal decongestants, clinically relevant nasal septum deviation, recurrent epistaxis) or sleep apnea;
* Elevated serum PSA levels (> 4 ng/ml for subjects >= 50 years of age);

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
The main study parameter is the change in sperm concentration during the 4-month study period for each of the two treatment groups. | 4 months

SECONDARY OUTCOMES:
The effects of treatment on the health related quality of life (QoL); | 4 months
The influence of transdermal and intranasal testosterone treatment on morphology and motility on sperm cells and on the volume of the ejaculate; | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Budumian, MD, Principal Investigator — AMPHA, Toernooiveld 220, 6525 EC Nijmegen, The Netherlands
Locations (1):
- AMPHA, Nijmegen, Netherlands